CLINICAL TRIAL: NCT07168538
Title: Effect of Transversus Abdominis Plane (TAP) Block on Postoperative Gastrointestinal Function After Laparoscopic Sleeve Gastrectomy: Evaluation Using the PRO-diGI Scale and Perlas Score (Prospective Clinical Study)
Brief Title: Effect of TAP Block on GI Function After Sleeve Gastrectomy Using PRO-diGI Scale and Perlas Score
Acronym: TAP
Status: Not yet recruiting | Type: Observational
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Sponsor
Other Study IDs: FSCH-SBÜ-2025/092
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Postoperative Gastrointestinal Dysfunction
Keywords: TAP Block; Gastrointestinal Motility; PRO-diGI Scale; Sleeve Gastrectomy
MeSH Terms: conditions — Obesity | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAP Block Group: Patients receiving bilateral ultrasound-guided TAP block at the end of laparoscopic sleeve gastrectomy as part of multimodal analgesia.
  Interventions: Procedure: TAP Block Group
- Control Group: Patients receiving standard multimodal analgesia without TAP block.
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: TAP Block Group — Bilateral ultrasound-guided transversus abdominis plane block performed at the end of surgery using 20 mL of 0.25% bupivacaine per side.
  Groups: TAP Block Group
Procedure: Control Group — Standard ERAS-based multimodal analgesia protocol without regional block.
  Groups: Control Group

SUMMARY:
This prospective clinical study aims to evaluate the effect of Transversus Abdominis Plane (TAP) block on postoperative gastrointestinal function in patients undergoing laparoscopic sleeve gastrectomy. Gastrointestinal recovery plays a crucial role in patient outcomes after bariatric surgery, and regional anesthesia techniques such as TAP block have been suggested to reduce postoperative pain and opioid consumption, which may influence gut motility.

In this study, postoperative gastrointestinal function will be assessed using the validated Patient-Reported Outcome for Dysfunctional Gastrointestinal Motility (PRO-diGI) scale. Additionally, gastric ultrasound will be performed to calculate the Perlas score as an objective marker of gastric emptying and residual volume. These assessments will allow a comprehensive evaluation of both subjective and objective gastrointestinal recovery parameters.

The study will include adult patients scheduled for elective laparoscopic sleeve gastrectomy at Elazığ Fethi Sekin City Hospital. Participants will receive standard general anesthesia with or without ultrasound-guided TAP block, and their postoperative recovery will be monitored. Primary outcomes include PRO-diGI scores at defined postoperative intervals, while secondary outcomes include Perlas scores obtained via gastric ultrasonography.

The findings from this research are expected to provide valuable insights into the potential benefits of TAP block on gastrointestinal motility and overall recovery after bariatric surgery.

DETAILED DESCRIPTION:
Bariatric surgery, particularly laparoscopic sleeve gastrectomy, is an effective intervention for morbid obesity. However, postoperative gastrointestinal dysfunction, including delayed gastric emptying and impaired gut motility, can adversely impact recovery, prolong hospital stay, and reduce patient satisfaction. Factors such as opioid-based analgesia are known contributors to postoperative ileus and gastrointestinal dysmotility. Therefore, optimizing pain management strategies while minimizing opioid use is critical for enhanced recovery.

The Transversus Abdominis Plane (TAP) block is a regional anesthesia technique that provides effective abdominal wall analgesia, reducing opioid consumption and associated adverse effects. While its role in postoperative pain control is well established, limited evidence exists regarding its impact on gastrointestinal function, particularly in the context of bariatric surgery.

Study Objective:

The primary objective of this study is to evaluate whether the application of ultrasound-guided TAP block affects postoperative gastrointestinal function after laparoscopic sleeve gastrectomy. Gastrointestinal recovery will be assessed using the PRO-diGI scale, which captures patient-reported symptoms of gastrointestinal motility, and the Perlas gastric ultrasound score, which provides an objective estimate of gastric content and residual volume.

Study Design:

This is a prospective, single-center clinical study conducted at Elazığ Fethi Sekin City Hospital. Adult patients scheduled for elective laparoscopic sleeve gastrectomy will be enrolled. All participants will receive standardized general anesthesia. TAP block will be administered as part of the perioperative analgesia strategy in eligible patients, based on clinical decision-making and patient consent.

Assessments:

Primary Outcome:

PRO-diGI score measured at predefined postoperative intervals (e.g., 6, 24, and 48 hours after surgery).

Secondary Outcomes:

Perlas score obtained via gastric ultrasonography in the early postoperative period.

Postoperative opioid consumption within the first 48 hours.

Incidence of postoperative nausea, vomiting, and ileus.

Length of hospital stay.

Ethics and Compliance:

The study will be conducted in accordance with the Declaration of Helsinki and Good Clinical Practice (GCP) guidelines. Ethical approval has been obtained from the institutional review board. Written informed consent will be obtained from all participants prior to study inclusion.

Expected Impact:

By integrating both subjective and objective measures of gastrointestinal function, this study will provide high-quality evidence regarding the potential benefits of TAP block beyond pain control. The results may contribute to optimizing perioperative care strategies for bariatric surgery and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-65 years
* Scheduled for primary laparoscopic sleeve gastrectomy (LSG)
* Body Mass Index (BMI) ≥ 35 kg/m²
* ASA Physical Status II-III
* Ability to provide written informed consent

Exclusion Criteria:

* Previous major abdominal surgery
* Known allergy to local anesthetics
* Severe hepatic or renal dysfunction
* Pregnancy or breastfeeding
* Conversion to open surgery during the procedure
* Patients refusing TAP block or general anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective laparoscopic sleeve gastrectomy at Elazığ Fethi Sekin City Hospital. Both male and female patients who meet inclusion criteria and consent to participate will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Gastrointestinal Function | Postoperative 6, 12, 24, and 48 hours
  Description: Assessed using the validated Patient-Reported Outcome for Dysfunction in Gastrointestinal Recovery after Surgery (PRO-diGI) scale, which captures patient-reported symptoms of gastrointestinal motility, including nausea, vomiting, bloating, and oral intake tolerance. The scale ranges from 0 to 15, with higher scores indicating greater gastrointestinal dysfunction and worse postoperative GI function.

SECONDARY OUTCOMES:
Perlas Score | Preoperative and immediate postoperative period
  Description: Gastric content and residual volume were assessed using bedside gastric ultrasound and graded according to the Perlas scoring system to estimate aspiration risk. Score 0 = empty antrum; Score 1 = minimal fluid in the right lateral decubitus; Score 2 = significant fluid in both supine and right lateral decubitus positions.
Opioid Consumption | First 48 hours postoperatively
  Total opioid use in morphine milligram equivalents.
Pain Scores (NRS) | 2, 6, 12, 24, and 48 hours postoperatively
  Patient-reported pain intensity measured using a numeric rating scale (NRS) from 0 (no pain) to 10 (worst possible pain) at rest and during movement. Higher scores indicate greater pain.
Adverse Events | From immediately after surgery up to 7 days postoperatively
  Incidence of postoperative nausea, vomiting, ileus, or TAP block-related complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided